CLINICAL TRIAL: NCT03532828
Title: Nocturnal Respiratory Disorders Identification and Their Influence on the Body Posture and Breathing Synchronisation in Patients With Dentofacial Dysgnathia
Brief Title: Interaction Between Body Posture and Nocturnal Sleeping Disorders in Dysgnathic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire de Biomécanique Georges Charpak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Dysmorphie / SAS
Record Dates: First submitted 2018-04-10; First posted 2018-05-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Dentofacial Deformities; Sleep Disorder; Posture
MeSH Terms: conditions — Dentofacial Deformities; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polysomnography alone (Experimental): A polygraphy will be performed in 70 patient to search for obstructive sleep apnea
  Interventions: Other: polysomnography
- Polysomnography and postural assesment (Experimental): A polygraphy and a postural assesment will be performed in 30 patients
  Interventions: Other: polysomnography

INTERVENTIONS:
Other: polysomnography — Patients will have a polygraphy, a postural evaluation including Vicon system, EOS imaging, ang a force platform
  Other Names: Postural evaluation

SUMMARY:
The role of head posture has been demonstrated in patient with dentofacial deformities. However, the relationship between body posture and jaw disorders is unclear. Moreover, patients with obstructive sleep apnea have the same anatomical abnormalities than patients with dentofacial deformities. The aim of this study is to evaluate, firstly, nocturnal sleeping disorders among patients with jaw disorders. Secondly, the investigators aim to evaluate the interaction between body posture, breathing and dentofacial deformities.

A polygraphy will be performed on patient with dentofacial deformities before and after correcting jaw surgery. A postural evaluation will be done using EOS imaging system and a force plate

ELIGIBILITY:
Inclusion Criteria:

* patient in orthodontic preparation for a surgical treatment,
* age > 16 years

Exclusion Criteria:

* postural disorder (scoliosis, history of spine surgery),
* pregnancy or breastfeeding,
* patients under guardianship

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in 2D displacement range of the pressure center | Baseline, 1 year
  Pressure center is recorded with force plates 1month before and 1 year after orthognathic surgery

SECONDARY OUTCOMES:
Change in EOS criteria description | Baseline, 1 year
  Criteria: pelvic tilt, cervical lordosis, C7 sagittal vertical axis, T1 slope thoracic kyphosis, lumbar lordosis , pelvic incidence, sacral slope. 1month before and 1 year after orthognathic surgery
Change Stabilometric criteria description | Baseline, 1 year
  2D displacement of the pressure center according to the anteroposterior axis, the lateral axis. 2D displacement speed. 1month before and 1 year after orthognathic surgery
Change in Cephalometric analysis | Baseline, 1 year
  Lateral cephalograms are recorded before and after surgery
Change Polygraphy criteria description | Baseline, 1 year
  Apnea-hypopnea index, oxygen saturation , before and after orthognathic surgery
Change in Dentofacial deformities description | Baseline, 1 year
  Clinical evaluation before and after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire de biomécanique Georges CHarpak, Paris, France

IPD SHARING:
Plan to Share IPD: No